CLINICAL TRIAL: NCT01328197
Title: A Phase I Clinical Study of the Safety and Performance of the Treovance Stent-Graft With Navitel Delivery System for Patients With Infrarenal Abdominal Aortic Aneurysms
Brief Title: Treovance Stent-Graft With Navitel Delivery System for Patients With Infrarenal Abdominal Aortic Aneurysms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0006-10
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Treovance; aneurysm; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Intervention Model Description: AAA device
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treovance (Experimental)
  Interventions: Device: Treovance Abdominal Aortic Stent-Graft with Navitel Delivery System

INTERVENTIONS:
Device: Treovance Abdominal Aortic Stent-Graft with Navitel Delivery System — Stent-graft implant

SUMMARY:
The primary goal of the study is to assess the safety and performance of the Treovance device in subjects with infrarenal aortic aneurysms, specifically to evaluate if the diseased pathology can be treated with an acceptable adverse event rate and that the device performs as expected. The results of this study will permit the establishment of endpoints and clinical design for a subsequent U.S. trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed with an infrarenal abdominal aortic aneurysm (AAA), with or without iliac artery involvement
* Subjects with an infrarenal AAA that is >/= 4.5 cm in diameter for males, or >/= 4.0 cm in diameter for females, or has increased in diameter by 0.5 cm in the last 6 months
* Subjects who consent to participate
* Subjects who agree to comply with the follow-up schedule

Exclusion Criteria:

* Subjects with dissections, ruptured aneurysms, or symptomatic aneurysms
* Subjects with prior AAA repair
* Subjects with medical conditions that would complicate the endovascular procedure or confound results (e.g., Marfan's syndrome, morbid obesity, severe coronary artery disease)
* Subjects who are pregnant or lactating
* Subjects participating in other investigational studies
* Subjects with less than 2 years life expectancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
major morbidity and mortality | 1, 6, 12 months

SECONDARY OUTCOMES:
Device performance | implant, 1, 6, and 12 months
  Rateof delivery/deployment success will be recorded. Rates of endoleak, patency, migration will be documented a 1, 6, 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Massachusetts, Worcester, Massachusetts
  - Spectrum Health System, Grand Rapids, Michigan
  - Carolinas Sanger Heart and Vascular, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sentara Heart Hospital, Norfolk, Virginia